CLINICAL TRIAL: NCT03698799
Title: Adherence Rate to Lung Protective Mechanical Ventilation in Patients Admitted to Surgical Intensive Care Units and Associated Clinical Outcomes
Brief Title: Adherence to LPV in SICU and Associated Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Annop Piriyapatsom, MD, Lecturer, Department of Anesthesiology, Principal Investigator, Mahidol University
Other Study IDs: 077/2561(EC4)
Record Dates: First submitted 2018-09-27; First posted 2018-10-09 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Adult; Guideline Adherence; Humans; Intensive Care Units; Perioperative/Postoperative Complications; Respiration, Artificial; Tidal Volume
Keywords: Adherence; Intensive Care Unit; Lung Protective Strategy; Mechanical Ventilation; Perioperative Critical Care; Surgical
MeSH Terms: conditions — Postoperative Complications; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LPV: Patients receive LPV strategy at the initiation of MV support. The LPV strategy is defined as ventilation with tidal volume of <8 mL/kg of PBW plus applying PEEP of at least 5 cm H2O.
- Non-LPV: Patients do not receive LPV strategy at the initiation of MV support.

SUMMARY:
Lung Protective Ventilation strategy (LPV) with low tidal volume and adequate positive end-expiratory pressure is recommended for not only patients with acute respiratory distress syndrome (ARDS) but also those without ARDS too. From previous studies, adherence to LPV strategy reported is only 40% and data is limited in surgical patients. The investigators aim to describe ventilation management and find out the adherence rate to LPV strategy applied to surgical patients admitted to the surgical intensive care unit (SICU) and their associated outcomes.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is one of the one organ support most frequently applied to patients admitted to intensive care units (ICUs). Despite considering as a life-saving intervention, MV may have detrimental effects, namely ventilator-induced lung injury (VILI). A mechanical breath with positive airway pressure may overstretch alveoli, especially in the non-dependent part of the lungs, and subsequently result in barotrauma and volutrauma. While cyclic opening and closing of alveoli during mechanical breath due to alveolar collapse at the end of expiration can cause atelec-trauma or cyclic atelectasis. All of these can lead to the activation of respiratory and systemic inflammatory response, so-called bio-trauma. To minimize the effects of MV on VILI, the lung protective mechanical ventilation (LPV) strategy have been proposed and now generally accepted as a standard practice in mechanically ventilated patients. The LPV strategy basically consists of ventilation with the low tidal volume of 6-8 mL/kg of predicted body weight (PBW) with limited plateau pressure of less than 30 cm H2O plus applying sufficient amount of positive end-expiratory pressure (PEEP) to prevent atelectasis. The LPV strategy has been clearly demonstrated benefits in not only patients with acute respiratory distress syndrome (ARDS) but also those with normal lungs including lessened respiratory and systemic inflammatory response and injured lungs, decreased duration of MV and length of stay (LOS), improved organ failure, and decreased pulmonary and other complications as well as mortality. Nevertheless, the adherence rate to the LPV strategy reported in the literatures is only approximately 40% in mechanically ventilated patients. For surgical patients, approximately 65% of those admitted to ICU require MV support either following operation or during their stay in ICU. To date, there is limited data regarding MV management in surgical patients who required MV support perioperatively. In addition, the difference in perioperative MV practices and their associated clinical outcomes has been not well determined in this setting. The aim of this study is to explore the current practice of MV according to the LPV strategy applied to surgical patients admitted to surgical ICU (SICU) and their associated clinical outcome. The primary outcome of this study is to determine the adherence rate to the LPV strategy at the initiation of MV support in mechanically ventilated patients in SICU. The LPV strategy in this study is defined as ventilation with the tidal volume of <8 mL/kg of PBW plus applying PEEP of at least 5 cm of water. The secondary outcomes are factors associated with the adherence to the LPV strategy, incidences of pulmonary and other complications, LOS in SICU and in hospital, SICU and hospital discharge status, and status at 28 and 90 days following the initiation of MV support. Patients are divided into two groups, LPV and Non-LPV, according to their MV setting and clinical outcomes are statistically compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age of 18 years old or more
* Patients admitted to two participating SICU
* Patients requiring MV support with the anticipated duration of 12 hours or more

Exclusion Criteria:

* Patients not requiring MV support during SICU stay
* Patients requiring MV support for less than 12 hours in SICU
* Patients requiring MV support for more than 24 hours prior to SICU admission
* Patients included in this study once and re-admitted to the SICU
* Patients requiring non-invasive MV support
* Moribund or terminal cases
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients whose age of 18 years old or more admitted to two participating SICU and requiring MV support, either at SICU admission or during stay in SICU, via either endotracheal or tracheostomy tube with the anticipated duration of 12 hours or more without exclusion criteria are included.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Adherence rate to LPV strategy at the initiation of MV support | During the first 24 hours following the initiation of MV support
  The LPV strategy is defined as ventilation with tidal volume of <8 mL/kg of PBW plus applying PEEP of at least 5 cm H2O.

SECONDARY OUTCOMES:
Incidences of pulmonary and other complications | During the first 7 consecutive days following the initiation of MV support
  Pulmonary complications include pneumonia, ARDS, atelectasis, restoration of MV support after liberation from MV, pleural effusion, cardiogenic pulmonary edema, pneumothorax and new pulmonary infiltration. Other complications include stroke, myocardial ischemia/infarction, arrhythmias, acute kidney injury, sepsis, new infection other than pneumonia, and re-admission to the SICU.
Length of stay in SICU and in hospital | Up to 90 days following the initiation of MV support
  Total days of stay in SICU and in hospital following the initiation of MV support.
SICU and hospital discharge status, and status at 28 and 90 days | Up to 90 days following the initiation of MV support
  Status whether alive or decease

CONTACTS AND LOCATIONS:
Overall Officials: Annop Piriyapatsom, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sutherasan Y, Vargas M, Pelosi P. Protective mechanical ventilation in the non-injured lung: review and meta-analysis. Crit Care. 2014 Mar 18;18(2):211. doi: 10.1186/cc13778. No abstract available. PMID 24762100
- [Background] Biehl M, Kashiouris MG, Gajic O. Ventilator-induced lung injury: minimizing its impact in patients with or at risk for ARDS. Respir Care. 2013 Jun;58(6):927-37. doi: 10.4187/respcare.02347. PMID 23709192
- [Background] Terragni P, Ranieri VM, Brazzi L. Novel approaches to minimize ventilator-induced lung injury. Curr Opin Crit Care. 2015 Feb;21(1):20-5. doi: 10.1097/MCC.0000000000000172. PMID 25546532
- [Background] Petrucci N, De Feo C. Lung protective ventilation strategy for the acute respiratory distress syndrome. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD003844. doi: 10.1002/14651858.CD003844.pub4. PMID 23450544
- [Background] Wang C, Wang X, Chi C, Guo L, Guo L, Zhao N, Wang W, Pi X, Sun B, Lian A, Shi J, Li E. Lung ventilation strategies for acute respiratory distress syndrome: a systematic review and network meta-analysis. Sci Rep. 2016 Mar 9;6:22855. doi: 10.1038/srep22855. PMID 26955891
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Neto AS, Simonis FD, Barbas CS, Biehl M, Determann RM, Elmer J, Friedman G, Gajic O, Goldstein JN, Linko R, Pinheiro de Oliveira R, Sundar S, Talmor D, Wolthuis EK, Gama de Abreu M, Pelosi P, Schultz MJ; PROtective Ventilation Network Investigators. Lung-Protective Ventilation With Low Tidal Volumes and the Occurrence of Pulmonary Complications in Patients Without Acute Respiratory Distress Syndrome: A Systematic Review and Individual Patient Data Analysis. Crit Care Med. 2015 Oct;43(10):2155-63. doi: 10.1097/CCM.0000000000001189. PMID 26181219
- [Result] Santamaria JD, Tobin AE, Reid DA. Do we practise low tidal-volume ventilation in the intensive care unit? a 14-year audit. Crit Care Resusc. 2015 Jun;17(2):108-12. PMID 26017128
- [Result] Kalhan R, Mikkelsen M, Dedhiya P, Christie J, Gaughan C, Lanken PN, Finkel B, Gallop R, Fuchs BD. Underuse of lung protective ventilation: analysis of potential factors to explain physician behavior. Crit Care Med. 2006 Feb;34(2):300-6. doi: 10.1097/01.ccm.0000198328.83571.4a. PMID 16424706
- [Result] Umoh NJ, Fan E, Mendez-Tellez PA, Sevransky JE, Dennison CR, Shanholtz C, Pronovost PJ, Needham DM. Patient and intensive care unit organizational factors associated with low tidal volume ventilation in acute lung injury. Crit Care Med. 2008 May;36(5):1463-8. doi: 10.1097/CCM.0b013e31816fc3d0. PMID 18434907
- [Result] Chen YF, Lim CK, Ruan SY, Jerng JS, Lin JW, Kuo PH, Wu HD, Yu CJ. Factors associated with adherence to low-tidal volume strategy for acute lung injury and acute respiratory distress syndrome and their impacts on outcomes: an observational study and propensity analysis. Minerva Anestesiol. 2014 Nov;80(11):1158-68. Epub 2014 Feb 25. PMID 24569355

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT03698799/Prot_SAP_000.pdf